CLINICAL TRIAL: NCT02945644
Title: Randomized Controlled Trial of Trazodone Dose Tolerance and APAP Adherence
Brief Title: Trazodone Dose Tolerance and APAP Adherence
Acronym: TrazoDose
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: COVID19 pandemic
Sponsor: Louis Stokes VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Kingman Strohl, Professor, Louis Stokes VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 16025-H17
Record Dates: First submitted 2016-10-11; First posted 2016-10-26 (Estimated); Last update posted 2020-05-11 (Actual); Status verified 2020-05

CONDITIONS: Sleep Apnea, Obstructive
Keywords: obstructive sleep apnea; trazodone; positive airway pressure; adherence
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Trazodone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo (Placebo Comparator): pill filled with inert material
  Interventions: Drug: Placebo
- Trazodone 50mg (Active Comparator)
  Interventions: Drug: Trazodone
- Trazodone 100mg (Active Comparator)
  Interventions: Drug: Trazodone

INTERVENTIONS:
Drug: Trazodone — take at bedtime for 14 days
  Other Names: oleptro; Desyrel
  Arms: Trazodone 100mg; Trazodone 50mg
Drug: Placebo — take at bedtime for 14 days
  Arms: Placebo

SUMMARY:
Trazodone may help obstructive sleep apnea patients to stick to their therapy, but optimal dosing is unknown. This study looks at what dose of trazodone has the best balance of potential benefits to side-effects in people with obstructive sleep apnea who are either starting on positive airway pressure therapy or not adherent to it. Participants will be randomly assigned to one of three groups: trazodone 50 mg, trazodone 100 mg, or placebo for 14 days. The investigators will monitor side-effects and adherence to positive airway pressure therapy.

DETAILED DESCRIPTION:
Clinical Significance: Trazodone is an often-used medication in clinical sleep medicine. However, there is a dearth of information on side-effects with doses typically used for sleep. In addition, a significant proportion of the VA population have obstructive sleep apnea for which the primary treatment is positive airway therapy. However, many patients have difficulty adhering to this treatment long-term. Increased adherence to this modality has been shown to improve risk for cardiovascular and neurologic co-morbidity associated with obstructive sleep apnea. This project explores both the tolerability and safety of common doses of trazodone used in clinical sleep practice as well explores potential effects on positive airway pressure therapy adherence.

Objectives: This project seeks to determine the tolerability and multi-domain effect on sleep and mood of a 14 day course of trazodone at either 50 mg or 100 mg or placebo.

Research Plan: This is a three-group, randomized, double-blind, placebo-controlled trial with prospective data collection of VA outpatient sleep clinic patients with obstructive sleep apnea with who are non-adherent or newly started on auto-titrating positive airway pressure therapy. Evaluation focuses on medication tolerability as measured by number of days before study drug discontinuation by the participant, the Treatment Satisfaction Questionnaire for Medication, the side-effect profile at the two doses (50mg and 100mg) compared to placebo as well as longitudinal collection of adherence data and standardized questionnaires on sleepiness, insomnia, depression, anxiety, and self-efficacy. The investigators also plan to longitudinally monitor coefficient of variation of breath-to-breath tidal volume, a measure of respiratory mechanics which may be affected by trazodone use. Study participants will have 2 visits at baseline and 2 weeks after randomization.

Methodology: This study will be conduced in the Louis Stokes Cleveland Medical Center - Wade Park Sleep Clinic, a tertiary institutional referral facility. Participants must be adults with obstructive sleep apnea prescribed auto-titrating positive airway therapy who are either newly initiated or do not fulfill standard criteria for adherence and do not have allergy to trazodone; current use of trazodone, monoamine oxidase inhibitors, or sedative hypnotics; alcohol or drug abuse; severe psychiatric disease; epilepsy; significant cardiac disease; liver disease; pregnancy; hypotension; or predisposition to priapism. Study staff will interview the potential participant and do a review of the medical record for exclusion criteria before consent is obtained. The investigators expect to recruit 45 participants into the study with a 20% attrition rate before completion. Hypothesis about the tolerability of trazodone and effect on positive airway therapy adherence was prespecified.

ELIGIBILITY:
Inclusion Criteria:

* Louis Stokes Cleveland VA Sleep Medicine clinic patient
* AHI greater than or equal to 5
* obstructive sleep apnea
* new initiation or nonadherence to APAP

Exclusion Criteria:

* schizophrenia
* bipolar disorder
* current use of trazodone or sedative hypnotics
* allergy to trazodone
* current use of tricyclic antidepressants or monoamine oxidase inhibitors
* current alcohol or drug abuse
* heart failure
* heart attack in past 3 months
* congenital long QT, ventricular arrhythmia (including Torsades de Pointes), bradycardia, or digoxin therapy
* use of amiodarone, sotalol, dofetilide, or dronedarone
* epilepsy
* liver disease
* pregnancy (or planning pregnancy)
* right of priapism: history of priapism, sickle cell disease, Farby disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2017-02-13 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Discontinuation rate by participant | 14-16 days post-randomization
  Did the participant discontinue trazodone at a higher rate than placebo?

SECONDARY OUTCOMES:
3 month APAP adherence | 3 months post-randomization assessing 30 days before this 3 month period
  APAP use in last 30 days (of the 3 month period) as measured by (1) average hours/day and (2) percent days with 4 or more hours use
Respiratory patterning | 14-16 days post-randomization
  Variation of breath to breath tidal volume obtained from plethysmography (a stretchy band around the chest x 20 minutes while wearing APAP)
Medication Satisfaction | 14-16 days post-randomization
  Treatment Satisfaction Questionnaire for Medications version II overall and subscale scores
side-effect profile | 14-16 days post-randomization
  participant-reported side effects of study drug
sleepiness | 14-16 days post-randomization
  Epworth Sleepiness Scale
insomnia | 14-16 days post-randomization
  Insomnia Severity Index
general self-efficacy | 14-16 days post-randomization
  General Self-Efficacy Scale
depression | 14-16 days post-randomization
  Clinically Useful Depression Outcome Scale (CUDOS)
anxiety | 14-16 days post-randomization
  Clinically Useful Anxiety Outcome Scale (CUXOS)

CONTACTS AND LOCATIONS:
Overall Officials: Kingman P Strohl, MD, Principal Investigator — Louis Stokes Cleveland VA Medical Center
Locations (1):
- Louis Stokes Cleveland VA Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No